CLINICAL TRIAL: NCT00415454
Title: Phase I Study Combining Replication-Competent Adenovirus-Mediated Suicide Gene Therapy With Chemoradiotherapy for the Treatment of Non-Metastatic Pancreatic Adenocarcinoma
Brief Title: Study Combining Suicide Gene Therapy With Chemoradiotherapy in the Treatment of Non-Metastatic Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Henry Ford Health System (Other)
Responsible Party: Svend O. Freytag, Ph.D., Henry Ford Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Panc4242; P01CA097012 (NIH)
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene therapy (Experimental): Adenovirus injection followed by 3 weeks of 5-FC + vGCV prodrug therapy and a 6 week course of capecitabine-based chemoradiation
  Interventions: Genetic: Ad5-yCD/mutTKSR39rep-ADP

INTERVENTIONS:
Genetic: Ad5-yCD/mutTKSR39rep-ADP — Single injection on day 1 at one of five dose levels

SUMMARY:
The primary purpose of this phase I study is to determine the safety of combining replication-competent adenovirus-mediated suicide gene therapy with chemoradiotherapy in patients with non-metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The objectives of this study are:

To determine the toxicity and maximum tolerated dose (MTD) of the Ad5-yCD/mutTKSR39rep-ADP adenovirus in combination with 5-fluorocytosine (5-FC) and valganciclovir (vGCV) prodrug therapy and standard chemoradiation. Fifteen to 30 subjects (5 cohorts of 3 - 6 subjects each) with non-metastatic, unresectable pancreatic cancer will receive a single intratumoral injection of the Ad5-yCD/mutTKSR39rep-ADP adenovirus at one of five dose levels (1 x 10e10 vp, 3 x 10e10 vp, 1 x 10e11 vp, 3 x 10e11 vp, 1 x 10e12 vp) under endoscopic ultrasound (EUS)-guidance. Beginning three days later, subjects will receive 3 weeks (15 days) of 5-FC and vGCV prodrug therapy concomitant with a 6 week (30 day) course of capecitabine chemotherapy and 54 Gy conformal radiotherapy.

The primary endpoint is toxicity at 12 weeks. Secondary endpoints are: 1) tumor (radiological) response, 2) time to disease progression, 3) survival, 4) persistence of Ad5-yCD/mutTKSR39rep-ADP adenoviral DNA in blood, 5) infectious Ad5-yCD/mutTKSR39rep-ADP adenovirus in blood, and 6) HSV-1 TK gene expression in the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 18 and < = 80.
* Non-metastatic, unresectable tumors
* No evidence of peritoneal and/or hematogenous metastasis.
* Histologically proven (biopsy or cytology) adenocarcinoma.
* No evidence of peritoneal and/or hematogenous metastasis.
* No prior chemotherapy, radiotherapy or biological therapy.
* ECOG performance status 0 - 2.
* Subjects must have adequate baseline organ function, as assessed by the following laboratory values, within 30 days before initiating the study therapy:
* Adequate renal function with serum creatinine <=1.5 mg/dL or creatinine clearance >=50 mL/min/m2.
* Absolute WBC > 4,000/μL.
* Hemoglobin > 9.0 g/dL.
* Platelet count > 100,000/μL.
* Bilirubin < 1.5 mg/dL; SGOT and SGPT < 2.5 times upper limit of normal (ULN).
* No history of malignancy within 5 years except for non-melanomatous skin cancer or carcinoma in situ of the cervix.
* Men and women with conceptive potential must agree to follow a medically acceptable method of birth control.
* Patients on oral warfarin anticoagulation therapy may be included in this study, but must have close monitoring of their coagulation parameters as altered parameters and/or bleeding have been reported in patients taking Xeloda® and such agents concomitantly.
* The subject must possess the ability to give informed consent and express a willingness to meet all of the expected requirements of the protocol for the duration of the study.

Exclusion Criteria:

* Pregnant and lactating women.
* Serious non-malignant disease (e.g., congestive heart failure or uncontrolled infections), which, in the opinion of the investigator would compromise study objectives.
* Major surgery within four weeks other than diagnostic procedures such as laparoscopy, endoscopic ultrasound and stenting or PEG/PEJ placement.
* Islet cell tumor, benign cyst, peri-ampullary carcinoma or any non-adenocarcinomas.
* Acute infection. Acute infection is defined by any viral, bacterial, or fungal infection that has required specific therapy within 72 hours of initiation of the study therapy (defined as Day 1).
* Active HIV disease.
* Previous history of liver disease including hepatitis.
* Positive serologic test for Hepatitis B or C at baseline.
* Immunosuppressive therapy including systemic corticosteroids. Use of inhaled and topical corticosteroids is permitted.
* Serious medical or psychiatric illness or concomitant medication, which, in the judgment of the investigator, might interfere with the subject's ability to respond to or tolerate the treatment or complete the trial.
* Impaired immunity or susceptibility to serious viral infections.
* Allergy to any product used on the protocol including ciprofloxacin.
* Clinical or laboratory evidence of pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Toxicity | 12 weeks post adenovirus injection

SECONDARY OUTCOMES:
Tumor response | 3 - 12 months
Time to progression | 3 - 12 months
Survival | 10 - 20 months
Gene expression in pancreas | 1 - 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Munther Ajlouni, M.D., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States